CLINICAL TRIAL: NCT02852993
Title: Survival After Blood Transfusion in the French Administrative Regions of Burgundy and Franche-Comté
Acronym: STeF-BFC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Centre Hospitalier Universitaire Dijon (Other); Etablissement Français du Sang (Other)
Responsible Party: Sponsor
Other Study IDs: P/2013/176
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Erythrocyte Transfusion for All Conditions
Keywords: Erythrocyte Transfusion; Survival

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Transfused patients: A cohort of patients receiving erythrocyte transfusion for the first time at the CHU Besançon or CHU Dijon during the study period.

SUMMARY:
Red blood cell transfusion (RBC) is the main symptomatic treatment for severe anemia. RBC transfusion has proven its efficacy regarding mortality and morbidity, but it is not without side effects. The infectious side effects of transfusion are largely considered under control, non-infectious side effects are taking center stage. Seeking explanations for the beneficial and deleterious effects of RBC transfusions is necessary to ensure the safe and optimal use of this precious resource.

The investigators aim to study the impact of donor and RBC characteristics on patient survival.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over
* Erythrocyte Transfusion between 2007 and 2011
* Performed at the University Hospital of Besançon or Dijon

Exclusion Criteria:

* Transfusion of any blood product prior to January 1st, 2007

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The eligible patients consisted of all adult patients transfused for the first time (defined as patients with no known history of RBC unit use in the transfusion register), at the university hospitals of Besançon or Dijon, between January 2007 and December 2011.
Sampling Method: Non-Probability Sample
Enrollment: 16099 (Actual)
Dates: Start 2013-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Desmarets, MD, PhD, Principal Investigator — Centre d'Investigation Clinique; CHU Besançon
Locations (2):
- France (2):
  - Centre d'Investigation Clinique, CHU de Besançon, Besançon
  - Département d'information Médicale, CHU Dijon, Dijon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Desmarets M, Bardiaux L, Benzenine E, Dussaucy A, Binda D, Tiberghien P, Quantin C, Monnet E. Effect of storage time and donor sex of transfused red blood cells on 1-year survival in patients undergoing cardiac surgery: an observational study. Transfusion. 2016 May;56(5):1213-22. doi: 10.1111/trf.13537. Epub 2016 Mar 2. PMID 26935140